CLINICAL TRIAL: NCT03259295
Title: Research on Current Prototypes of the Digiclamp. Short Term and Long Term Outcomes of Treating Adults With Achrocordons (Skin Tags)
Brief Title: Study to Evaluate the Efficacy of Removing Skin Tags With Digiclamp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: XDG Technologies, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20171314 - WIRB; PRO00002692 (Other: University of Florida Project #)
Record Dates: First submitted 2017-08-21; First posted 2017-08-23 (Actual); Results first posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Achrochordon
Keywords: skin tag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Skin tag removal initial visit plus follow-up (Experimental): Removal of skin tags 1 cm or less using Digiclamp and follow-up 2-3 months after skin tag removal to assess functionality and effectiveness of the device.
  Interventions: Device: Digiclamp (Skin tag removal initial plus follow-up)

INTERVENTIONS:
Device: Digiclamp (Skin tag removal initial plus follow-up) — Skin tag will be assessed for size, location, and overall appearance. After assessment and confirmation that the skin tag is not infected or possibly malignant, the site will be photographed, prepped with an antimicrobial solution, anesthetized, and removed using the Digiclamp. A bandaid will be applied to the site. Site of skin tag removal will be photographed to document lesion recurrence and presence of scar tissue or hyperpigmentation. Subjects will be asked to complete a brief survey about their satisfaction with the use of Digiclamp.

SUMMARY:
The objective of this study is to assess the efficacy of using the Digiclamp device to remove achrocordons (skin tags). The hypothesis is that utilizing the device will result in low rates of re-occurrence, scars, scar tissue and discoloration at the site of removal.

DETAILED DESCRIPTION:
Achrocorodons, or skin tags, are superficial cutaneous lesions that occur most commonly among middle aged adults, obese persons and those who suffer from Type 2 Diabetes. In most cases, the tags are not bothersome but there are instances when they can become infected or irritated. There are several skin tag removal options available, including suture ligature, freezing, cautery or excision. These procedures are often done in a dermatology office and are an out-of-pocket cost.

The Digiclamp device was invented to make skin tag removal procedures more accessible. The Digiclamp represents a new option that when placed in the hands of primary care clinicians, it will allow them to remove skin tags without having to purchase expensive devices or to refer them to a Dermatologist. The device is disposable, and relatively painless when used correctly, and requires minimal training.

The investigator is planning to enroll 100 subjects, who will have skin tags removed using the Digiclamp device. Subjects will return for follow up at 2-3 months after skin tag removal.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with simple skin tag(s) measuring up to 1 centimeter width at the base of the skin tag

Exclusion Criteria:

* Subjects with skin tags measuring greater than 1 centimeter width at the base
* Subjects whose skin tags appear infected or may need to be evaluated by pathology
* Subjects whose skin tags are located in genital areas or eyelids
* Pregnant subjects
* Subjects with bleeding disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan C Roig, MD, Principal Investigator — University of Florida
Locations (1):
- Office of Raymond Marquette, MD, Ocala, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Watson BT, Hennrikus WL. Postaxial type-B polydactyly. Prevalence and treatment. J Bone Joint Surg Am. 1997 Jan;79(1):65-8. doi: 10.2106/00004623-199701000-00007. PMID 9010187
- [Background] Schmook T, Stockfleth E. Current treatment patterns in non-melanoma skin cancer across Europe. J Dermatolog Treat. 2003;14 Suppl 3:3-10. doi: 10.1080/jdt.14.s3.3.10. PMID 14522635
- [Background] Kahana M, Grossman E, Feinstein A, Ronnen M, Cohen M, Millet MS. Skin tags: a cutaneous marker for diabetes mellitus. Acta Derm Venereol. 1987;67(2):175-7. PMID 2438887
- [Background] Banik R, Lubach D. Skin tags: localization and frequencies according to sex and age. Dermatologica. 1987;174(4):180-3. doi: 10.1159/000249169. PMID 3582706

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Skin Tag Removal Initial Visit Plus Follow-up
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Skin Tag Removal Initial Visit Plus Follow-up
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (9.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Weight [Mean (Standard Deviation); unit: pounds] | 182 (43.9)
Height [Mean (Standard Deviation); unit: inches] | 66.4 (3.07)
Number of lesions [Mean (Standard Deviation); unit: lesions] | 2.5 (1.15)
Location of lesions [Number; unit: lesions]
  neck | 19
  maxilla | 1
  axilla | 7
  back | 8
  areola | 1
  thigh | 2
  rib cage | 1
  buttock | 1
  mandible | 2
  shoulder | 2
  abdomen | 2
  chest | 4
width of lesion [Mean (Standard Deviation); unit: cm] | 0.404 (0.276)
height of lesion [Mean (Standard Deviation); unit: cm] | 0.376 (0.252)

OUTCOME MEASURES:

1. Primary Outcome: Re-occurrence Rate of Skin Tags
Description: Percentage of subjects who experience a re-occurrence of the skin tag at the removal site.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Skin Tag Removal Initial Visit Plus Follow-up
Number analyzed (Participants) | 20
Participants | 0

2. Secondary Outcome: Percentage of Permanent Scars Among Lesion Sites
Description: Percentage of subjects who develop a scar at the removal site
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Skin Tag Removal Initial Visit Plus Follow-up
Number analyzed (Participants) | 20
Participants | 1

3. Secondary Outcome: Percentage of Scar Tissue Formation Among Lesion Sites
Description: Percentage of subjects who develop scar tissue or keloid at the site of removal
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Skin Tag Removal Initial Visit Plus Follow-up
Number analyzed (Participants) | 20
Participants | 0

4. Secondary Outcome: Percentage of Discoloration Among Subjects
Description: Percentage of subjects who develop discoloration at the site of removal
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Skin Tag Removal Initial Visit Plus Follow-up
Number analyzed (Participants) | 20
Participants | 3

5. Secondary Outcome: Percentage of Pain/Numbness Where Skin Tag Was Removed
Description: Percentage of subjects who develop pain/numbness at the site of removal
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Skin Tag Removal Initial Visit Plus Follow-up
Number analyzed (Participants) | 20
Participants | 0

6. Secondary Outcome: Satisfaction With Pain Post Procedure
Description: All study participants were asked three questions in a post procedure satisfaction survey.
  1. How satisfied are you with the amount of pain you experienced while having your skin tag removed? Study participants responded whether they were "very satisfied", "somewhat satisfied", "neither satisfied nor dissatisfied", "somewhat dissatisfied", "very dissatisfied". Subjects were counted in each category and reported.
Time Frame: 2 months post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Skin Tag Removal Initial Visit Plus Follow-up
Number analyzed (Participants) | 20
Participants
  Very satisfied | 20
  Somewhat satisfied | 0
  Neither satisfied nor dissatisfied | 0
  Somewhat dissatisfied | 0
  Very dissatisfied | 0

7. Secondary Outcome: Satisfaction With What the Area Looked Like Post Procedure
Description: All study participants were given a satisfaction survey 2 months post procedure. Subjects had to choose if they were "very satisfied:, "somewhat satisfied", "neither satisfied nor dissatisfied", "somewhat dissatisfied", "very dissatisfied" with how the area looks where the skin tag used to be. Subjects in each category were counted and reported.
Time Frame: 2 months post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Skin Tag Removal Initial Visit Plus Follow-up
Number analyzed (Participants) | 20
Participants
  Very satisfied with how the area looked like where the skin tag used to be | 19
  Somewhat satisfied with what the area looked like | 1
  Neither satisfied nor dissatisfied | 0
  Somewhat dissatisfied | 0
  Very dissatisfied | 0

8. Secondary Outcome: How Likely to Recommend the Procedure to Friends and Family
Description: All study participants were asked a satisfaction survey post procedure and whether they would recommend the procedure to friends and family. Categories for response were: "very likely", "somewhat likely", "neither likely nor unlikely", "somewhat unlikely", "very unlikely". Subjects in each category were counted and reported.
Time Frame: 2 months post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Skin Tag Removal Initial Visit Plus Follow-up
Number analyzed (Participants) | 20
Participants
  Very likely to recommend the procedure to friends and family | 20
  Somewhat likely | 0
  Neither likely nor unlikely | 0
  Somewhat unlikely | 0
  Very unlikely | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Skin Tag Removal Initial Visit Plus Follow-up
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2017-07-17): https://cdn.clinicaltrials.gov/large-docs/95/NCT03259295/Prot_002.pdf